CLINICAL TRIAL: NCT05884931
Title: A Prospective, Multicenter, Open-label, Randomized Controlled Study to Evaluate Safety and Effectiveness of Endoscopic Hemostatic Powder, 'Nexpowder' for Hemostatic Treatments of Lower Gastrointestinal Bleeding After Colon Polypectomy
Brief Title: Effectiveness and Safety of Nexpowder as an Endoscopic Hemostatic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nexpowder_02
Record Dates: First submitted 2023-05-08; First posted 2023-06-01 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: GastroIntestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (Active Comparator): Conventional Treatment
  Interventions: Procedure: Conventional Treatment
- Conventional Treatment + Nexpowder (Experimental): Conventional Treatment + Nexpowder
  Interventions: Device: Nexpowder

INTERVENTIONS:
Device: Nexpowder — Hemostatic powder for endoscopy after colonoscopy polypectomy
  Arms: Conventional Treatment + Nexpowder
Procedure: Conventional Treatment — Standard hemostatic procedure
  Arms: Conventional Treatment

SUMMARY:
In patients who show signs of bleeding and bleeding after polypectomy such as EMR and ESD for polyps with a diameter of 2 cm or more in the lower gastrointestinal tract, the effectiveness and safety of Nexpowder as an endoscopic hemostatic treatment are confirmed.

DETAILED DESCRIPTION:
Total number of target subjects 66 Test group 33 / Control group: 33 If endoscopic polypectomy is performed on polyps of 2cm or more, the probability of bleeding as a complication is 6.5%. This clinical study is an observational study to confirm the safety and effectiveness of Nexpowder, an endoscopic hemostatic powder after colonoscopy polypectomy, and an exploratory evaluation of 60 patients is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Adult volunteers aged 19 or older during screening
2. A person who is scheduled to perform polypectomy for polyps with a diameter of 2 cm or more, such as Endoscopic Mucosal Resection (EMR) or Endoscopic Submucosal Dissection (ESD)
3. If the researcher agrees to voluntarily participate in the clinical study and determines that the subject cannot voluntarily consent due to the elderly aged 80 or older or other emergency situations, a written consent of the subject's legal representative is required

Exclusion Criteria:

1. Upper gastrointestinal bleeding
2. If ulcerative bleeding is not caused by the procedure
3. If you are suffering from a blood clotting disorder
4. Aspirin and anticoagulant medications cannot be discontinued
5. Pregnant or lactating
6. Where colonoscopy is prohibited due to comorbid diseases, etc
7. If the bleeding area cannot be identified or the bleeding area cannot be reached with an endoscope
8. If you have participated in a relevant clinical trial that may affect the results of this study within the last one month
9. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose galactose malabsorption
10. A person who is hypersensitive to food additive Blue No. 1 or has a history of allergies
11. In the case where the researcher determines that it is inappropriate to participate in clinical trials due to other reasons other than the above selection exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Rate of rebleeding within 7 days of successful endoscopic hemostasis | 7 days
  Rate of rebleeding within 7 days of successful endoscopic hemostasis
Rate of rebleeding within 30 days of successful endoscopic hemostasis Except for cases of rebleeding within 7 days of successful endoscopic hemostasis) | 30 days
  Rate of rebleeding within 30 days of successful endoscopic hemostasis Except for cases of rebleeding within 7 days of successful endoscopic hemostasis)

SECONDARY OUTCOMES:
Check for haemostasis within 5 minutes from the moment of application of Nexpowder Analysis of patients with bleeding during the initial hemostasis experimental group | 5 min
  Check for haemostasis within 5 minutes from the moment of application of Nexpowder Analysis of patients with bleeding during the initial hemostasis experimental group
Perforation incidence | 7 days
  Perforation incidence
Death rate | 7 days
  Death rate
Blood transfusion case rate | 7 days
  Blood transfusion case rate
Number of Nexpowder applications (experimental group) | 7 days
  Number of Nexpowder applications (experimental group)
Number of usage of Nexpowder (experimental group) | 7 days
  Number of usage of Nexpowder (experimental group)
Incidence of device malfunction (experimental group) | 7 days
  Incidence of device malfunction (experimental group)
Rate of ease of use (experimental group) | 7 days
  Rate of ease of use (experimental group)

OTHER OUTCOMES:
Abnormal response intestinal obstruction, including gas embolism during a 30-day follow-up period | 30 days
  Abnormal response intestinal obstruction, including gas embolism during a 30-day follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Kibae Kim, Ph.D., Study Director — Chungbuk National University Hospital
Locations (3):
- South Korea (3):
  - Chungbuk National University Hospital, Cheongju-si
  - Chungnam National University Hospital, Daejeon
  - Chungnam National University Sejong Hospital, Sejong

IPD SHARING:
Plan to Share IPD: No